CLINICAL TRIAL: NCT04375774
Title: Verification of Alternative Do-it-yourself Equipment Respirators
Brief Title: Verification of Alternative Do-it-yourself Equipment Respirators for the COVID-19 Personal Protective Equipment (PPE)
Acronym: VADER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020/15AVR/226
Record Dates: First submitted 2020-04-17; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: COVID
Keywords: COVID; protection equipment; 3d printable valve; fit test

STUDY DESIGN:
Intervention Model Description: Enrolment will be a onetime selection of 10 healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FFP2 (Other)
  Interventions: Device: FFP2
- Facial mask (Other)
  Interventions: Device: Facial mask
- Modified full-face snorkeling (Other)
  Interventions: Device: MFS

INTERVENTIONS:
Device: FFP2 — Face Fit test of the FFP2 with the PortaCount® PRO+ 8038 from TSI
  Arms: FFP2
Device: Facial mask — Face Fit test of a conventional respirator facial mask with the PortaCount® PRO+ 8038 from TSI
  Arms: Facial mask
Device: MFS — Face fit test of a MFS with the PortaCount® PRO+ 8038 from TSI
  Arms: Modified full-face snorkeling

SUMMARY:
The COVID-19 pandemic health crisis forces health institutions to lower their standards of protection as supplies of personal protective equipment decrease despite the safety of front-line workers worldwide . This shortage specifically affects high-quality protective masks, such as those called FFP2. As alternatives, we offer a reusable mask based on a ventilation mask combined with a breathing filter for anesthesia breathing circuits. The purpose of the study is to assess the sealing potential of this mask in the field and possibly prove a non-inferior sealing compared to standard masks type FFP2.

DETAILED DESCRIPTION:
The ongoing 2020 COVID-19 pandemic challenges healthcare providers (HCP) worldwide with a rapid consumption and shortage of personal protection equipment (PPE), especially high-level filtration respirator masks. Respirators used by HCPs are mainly single use face filtering pieces with at least level P2 protection for single shift use following European EN 149 standards defining protection level against hazardous particles.

In response to the risk of shortage we propose a novel reusable do-it-yourself (DIY) respirator assembled with already widely available components in hospital stocks: a standard breathing filter plugged in an anaesthesia facial mask held in place with a hook ring strapped to a silicone head harness. As reports of a modified full-face snorkelling (MFS) mask used for non-invasive ventilation in infected patients emerged in Italy, we reckon that it could also be used as PPE with a modified valve and breathing filter.

ELIGIBILITY:
Inclusion Criteria:

* adult volunteers working in a first line healthcare service with basic knowledge of donning PPE including respirators
* 5 females and 5 males

Exclusion Criteria:

* smoking or unhealthy participants with respiratory affections to avoid breathing difficulties during testing
* any known allergy towards medical silicone or any other material of each component and ingredients used for disinfection of the test area and material between participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of airtightness (Fit test) | Up to 1 week
  Non inferiority claim over FFP2

SECONDARY OUTCOMES:
User Comfort | Up to 1 week
  User face comfort for each type of mask assessed by a assessed by a scoring-cale from 1 to 5
Breathing easiness | Up to 1 week
  User respiratory easiness for each type of mask assessed by a scoring-cale from 1 to 5
Field of view quality | Up to 1 week
  User field of view quality for each type of mask assessed by a scoring-cale from 1 to 5
Ease of use | Up to 1 week
  How the device is user friendly, assessed by a scoring-cale from 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lemaire, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
All data will be presented in the future manuscript